CLINICAL TRIAL: NCT04738825
Title: Promoting HIV Risk Reduction Among People Who Inject Drugs: A Stepped Care Approach Using Contingency Management With PrEP Adherence and Support Services
Acronym: CoMPASS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000029351; R01DA051871 (NIH)
Record Dates: First submitted 2021-01-29; First posted 2021-02-04 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Opioid-use Disorder; HIV Prevention Program
Keywords: People who inject drugs; Pre-exposure prophylaxis (PrEP); Medications for opioid use disorder; Opioid use disorder; HIV prevention
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Aims 1 and 2: Randomized controlled trial to evaluate the effectiveness of contingency management with stepped care to PrEP adherence and support services (Compass) compared to treatment as usual.
  Aim 3: Implementation-focused process evaluation to gain information on implementation of the intervention from perspectives of participants as well as front-line providers and staff
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (TAU) (No Intervention): Participants randomized to TAU will receive a health handout on HIV risk reduction approaches, including PrEP and OUD-related care, and where to access such services. They will receive standard care as provided by the community-based organization and by their medical provider.
- Contingency Management with stepped care to PrEP Adherence and Support Services (CoMPASS) (Experimental): Participants randomized to Compass will also receive a health handout on HIV risk reduction approaches. They will also receive contingency management sessions (n=9). Participants who do not demonstrate PrEP adherence by week 12, will be "stepped up" to receive PrEP adherence and support services (n=5).
  Interventions: Behavioral: Contingency Management with stepped care to PrEP adherence and support services (CoMPASS)

INTERVENTIONS:
Behavioral: Contingency Management with stepped care to PrEP adherence and support services (CoMPASS) — Participants will receive contingency management sessions (n=9). Participants who do not demonstrate PrEP adherence by week 12 will be "stepped up" to receive PrEP adherence and support services (n=5).
  Arms: Contingency Management with stepped care to PrEP Adherence and Support Services (CoMPASS)

SUMMARY:
The proposed study will be a 24-week intervention with a 12-month follow-up period to evaluate the impact of contingency management with stepped care to pre-exposure prophylaxis (PrEP) adherence and support services (CoMPASS) to promote HIV prevention among individuals with opioid use disorder who have injected drugs in their lifetime. In parallel, the investigators will conduct an implementation focused process evaluation to inform real-world implementation of CoMPASS. .

DETAILED DESCRIPTION:
Consistent with a Hybrid Effectiveness-Implementation Type 1 design, this is a multi-site randomized clinical trial designed to evaluate the effectiveness of Contingency Management with stepped care to PrEP Adherence and Support Services (CoMPASS) vs. treatment as usual (TAU) on HIV risk reduction among individuals with opioid use disorder (OUD) who have injected drugs in their lifetime. The study will be conducted in community-based settings serving individuals with opioid use disorder to assess the effectiveness of CoMPASS on promoting: sustained PrEP adherence (primary outcome) and HIV risk behaviors, engagement in opioid use disorder-related care, opioid use (secondary outcomes); and sexually transmitted infections and HIV (exploratory). Participants randomized to CoMPASS will first receive contingency management and have the potential to earn prizes for making progress towards initiation of and consistent adherence to HIV pre-exposure prophylaxis (PrEP) and engagement in OUD-related care. Individuals who do not demonstrate PrEP adherence (based on self-report, confirmed by urine testing for tenofovir metabolites at week 12), will be "stepped up" to PrEP Adherence and Support Services (PASS). The intervention is 24 weeks in duration. Participants randomized to TAU will receive a health handout on HIV risk reduction approaches, including PrEP and OUD-related care, and where to access such services.

To inform future implementation efforts, factors relevant for scale-up in parallel (e.g., completion of study visits, attitudes regarding the intervention among front-line staff) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Aims 1 and 2:

1. Receive or willing to receive care at one of the participating study sites
2. Have a recent negative HIV test with no concern for acute HIV
3. Report injection drug use in their lifetime
4. Meet PrEP eligibility criteria by either a) sharing of injection or drug preparation equipment; b) sexual risk behaviors (i.e. condomless sex or STI) in the past 6 months
5. Meet Diagnostic and Statistical Manual of Mental Disorders - 5th edition (DSM5) criteria for opioid use disorder
6. Have a phone or use of a household member's phone
7. Provide written informed consent

Aim 3:

1. Currently employed at one of the participating study sites
2. Willing to complete a web-based survey

Exclusion criteria:

Aims 1 and 2:

1. Currently prescribed PrEP
2. Self-report or urine test confirming pregnancy, breastfeeding, or trying to conceive
3. Any plans that would preclude study completion (surgery, major medical treatment or conditions, incarceration, travel out of state or country.)
4. Inability to provide at least one collateral contact for a friend or family member.
5. Non-English speaking (for sites without Spanish-speaking staff)
6. Have kidney disease (a contraindication to PrEP)

Aim 3:

1. Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sustained PrEP adherence | 24 weeks
  Determined by tenovifir-diphosphate levels by dried blood spot testing.

SECONDARY OUTCOMES:
Sustained PrEP adherence | 12 weeks
  Determined by tenovifir-diphosphate levels by dried blood spot testing. .
Recent PrEP adherence | 12 weeks
  Self-report adherence confirmed by the presence of tenofivir in urine sample.
HIV Risk Behaviors | 12 weeks
  Self-reported HIV risk behaviors
HIV Risk Behaviors | 24 weeks
  Self-reported HIV risk behaviors
Engagement in opioid use disorder-related care | 12 weeks
  Self report of engagement in opioid use disorder-related care
Engagement in opioid use disorder-related care | 24 weeks
  Self report of engagement in opioid use disorder-related care
Extra medical opioid use | 12 weeks
  Self reported extra medical opioid use
Extra medical opioid use | 24 weeks
  Self reported extra medical opioid use

OTHER OUTCOMES:
Sexually transmitted infection and HIV acquisition | 12 months
  State surveillance data

CONTACTS AND LOCATIONS:
Overall Officials: E. Jennifer Edelman, MD, MHS, Principal Investigator — Yale University
Locations (6):
- United States (6):
  - Recovery Network of Programs, Inc, Bridgeport, Connecticut
  - Liberations Program, Inc, Bridgeport, Connecticut
  - Apex Community Care. Inc., Danbury, Connecticut
  - Greater Hartford Harm Reduction Coalition- SWAN, New Haven, Connecticut
  - APT, New Haven, Connecticut
  - Stanley Street Treatment and Resource Center, Fall River, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pickering E, Viera A, Sung ML, Davidson D, Bailey G, Buchelli M, Jenkins M, Kolakowski J, Maier L, Edelman EJ, Rash CJ. Readiness to implement contingency management to promote PrEP initiation and adherence among people who inject drugs: results from a multi-site implementation survey. Addict Sci Clin Pract. 2024 Dec 23;19(1):97. doi: 10.1186/s13722-024-00503-4. PMID 39710733
- [Derived] Sung ML, Viera A, Esserman D, Tong G, Davidson D, Aiudi S, Bailey GL, Buchanan AL, Buchelli M, Jenkins M, John B, Kolakowski J, Lame A, Murphy SM, Porter E, Simone L, Paris M, Rash CJ, Edelman EJ. Contingency Management and Pre-Exposure Prophylaxis Adherence Support Services (CoMPASS): A hybrid type 1 effectiveness-implementation study to promote HIV risk reduction among people who inject drugs. Contemp Clin Trials. 2023 Feb;125:107037. doi: 10.1016/j.cct.2022.107037. Epub 2022 Nov 30. PMID 36460267